CLINICAL TRIAL: NCT01550263
Title: Pre-Operative Psychological Distress and Post-Operative Outcomes in Hip Preservation Patients
Brief Title: Psychological Distress and Outcomes in Hip Preservation Patients
Acronym: Hip
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Stephen Aoki, M.D., University of Utah
Other Study IDs: 48948
Record Dates: First submitted 2012-02-08; First posted 2012-03-09 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Psychological Distress
Keywords: Hip Preservation; Hip Arthroscopy; Hip Pain; Psychological distress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an investigatory study to determine whether high levels of pre-operative psychological distress predict worse outcomes after hip preservation. This is a low risk study and does not alter the treatment or course of care for patients undergoing this procedure

DETAILED DESCRIPTION:
The correlation between increasing psychological distress and worsening surgical outcomes has been extensively documented in patients undergoing spine surgery. However, we have no reason to believe that patients with hip pathology are uniquely exempt from the influence of psychosocial factors. To our knowledge, no study has been done to evaluate the effect of pre-operative psychological distress on outcomes after hip preservation surgery. We therefore propose to use the DRAM to measure pre-operative distress in patients undergoing open or arthroscopic hip preservation surgery and to compare these pre-operative distress scores with post-operative outcomes. We hope the information we gain will allow clinicians to comprehensively evaluate the patient with hip pain and to make more informed choices about operative treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Primary presenting complaint of hip pain
2. Hip arthroscopy, surgical dislocation and debridement, and/or periacetabular osteotomy performed by Dr. Aoki or Dr. Peters for hip pathology diagnosed by history, clinical examination and/or imaging

Exclusion Criteria:

1. Unable to complete the DRAM questionnaire
2. Patients who do not undergo surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are selected by Dr. Aoki
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2012-01; Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Distress and Risk Assessment Method (DRAM) questionaire | 1 year
  Distress and Risk Assessment Method (DRAM) questionaire to screen for psychological distress. The instrument defines four categories based on patients responses: Type N (normal; lower scores, no evidence of distress); Type R (at risk; higher scores, primarily in symptoms of depression); Type DD (distressed-depressive; higher scores on all variables, but very high on depressive symptomatology); and Type DS (distressed-somatic; higher scores on all variables, but very high on somatic awareness).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen K Aoki, MD, Principal Investigator — Orthopaedic Center
Locations (1):
- Orthopaedic Center, Salt Lake City, Utah, United States